CLINICAL TRIAL: NCT00006228
Title: Phase II Trial of Anti-HER-2 Monoclonal Antibody Trastuzumab (Herceptin) in Combination With Low Dose Interleukin-2 (Proleukin) in Metastatic Breast Cancer Patients Who Have Previously Failed Trastuzumab
Brief Title: Trastuzumab and Interleukin-2 in Treating Patients With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01402; NCI-2012-01402 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000068150; OSU-99H0192; OSU-9945; NCI-195; 9945 (Other: Ohio State University Medical Center); 195 (Other: CTEP); N01CM17102 (NIH)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2013-10-08 (Estimated); Status verified 2013-10

CONDITIONS: HER2-positive Breast Cancer; Male Breast Cancer; Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms, Male; Breast Neoplasms | interventions — Trastuzumab; aldesleukin

ARMS (1):
- Treatment (trastuzumab and aldesleukin) (Experimental): Patients receive trastuzumab IV over 30-90 minutes on days 1 and 8 and aldesleukin SC on days 2-7 and 9-21. Beginning on day 22, patients receive trastuzumab IV over 30 minutes every 14 days. Patients also receive aldesleukin SC daily on days 1-14. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: trastuzumab; Biological: aldesleukin; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Biological: trastuzumab — Given IV
Biological: aldesleukin — Given SC
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies

SUMMARY:
Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Interleukin-2 may stimulate a person's white blood cells to kill breast cancer cells. Phase II trial to study the effectiveness of trastuzumab plus interleukin-2 in treating patients who have metastatic breast cancer that has not responded to previous trastuzumab therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the response rate and toxicity to low-dose IL-2 with intermediate-"pulse" dose interleukin 2 (IL-2) and trastuzumab in patients with uni-dimensional measurable metastatic breast cancer and human epidermal growth factor receptor 2 (HER2) positive (3+ overexpression by immunohistochemistry [IHC] method or positive by fluorescent in situ hybridization [FISH]) who either have had evidence of progressive disease while receiving a trastuzumab-containing regimen, or have had progressive disease within 12 months of receiving a trastuzumab-containing regimen.

SECONDARY OBJECTIVES:

I. To perform correlative immunologic assays to determine the degree of natural killer (NK) cell expansion in response to low-dose IL-2, and the effectiveness of patients' peripheral blood mononuclear cells (PBMC) in a standard antibody-dependent cell-mediated cytotoxicity (ADCC) assay directed against a HER2 target cell.

II. To determine the pharmacokinetics of trastuzumab using an every 2-week schedule.

III. To determine Fc-gamma receptor polymorphisms from study patients.

OUTLINE: This is a multicenter study.

Patients receive trastuzumab intravenously (IV) over 30-90 minutes on days 1 and 8 and aldesleukin subcutaneously (SC) on days 2-7 and 9-21. Beginning on day 22, patients receive trastuzumab IV over 30 minutes every 14 days. Patients also receive aldesleukin SC daily on days 1-14. Treatment continues for 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days.

PROJECTED ACCRUAL: A total of 17-37 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed breast cancer

  * Primary and/or metastatic disease
* HER2 overexpression 3+ by immunohistochemistry (IHC) or fluorescence in situ hybridization (FISH)

  * Tumors with HER2 2+ overexpression by IHC allowed if confirmed by FISH
* Progressive disease during or within 12 months of receiving prior regimen containing trastuzumab (Herceptin)
* Unidimensionally measurable disease

  * At least 20 mm by conventional techniques OR at least 10 mm by spiral CT scan
  * The following are not considered measurable:

    * Bone metastases
    * Pleural or peritoneal effusion
    * Ascites
    * Leptomeningeal disease
    * Lymphangitic disease
    * Inflammatory breast cancer
    * Cystic lesions
    * CNS lesions
* CNS metastases allowed if all of the following conditions are met:

  * Asymptomatic
  * At least 3 months since prior surgery and/or cranial irradiation
  * At least 3 weeks since prior steroids
* Hormone receptor status:

  * Not specified
* Male or female
* Performance status - ECOG 0-2
* Granulocyte count at least 1,000/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2 times ULN (5 times ULN for liver metastases)
* Alkaline phosphatase no greater than 2 times ULN (5 times ULN for liver metastases)
* Creatinine no greater than 1.5 times ULN
* LVEF at least lower limit of normal by MUGA or echocardiogram
* No congestive heart failure or active ischemic heart disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No psychiatric illness, medical condition, or uncontrolled infection that would preclude study
* No underlying immunodeficiency (e.g., HIV or autoimmune disease)
* No other prior malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* See Disease Characteristics
* Prior cumulative doxorubicin dose no greater than 360 mg/m^2
* At least 3 weeks since prior chemotherapy
* No more than 2 prior chemotherapy regimens for metastatic disease
* No concurrent chemotherapy
* See Disease Characteristics
* At least 3 weeks since prior endocrine therapy
* No concurrent corticosteroids or dexamethasone
* Concurrent hormones allowed for conditions unrelated to disease (e.g., insulin for diabetes)
* See Disease Characteristics
* At least 3 weeks since prior radiotherapy
* No prior radiotherapy to study lesion, unless evidence of disease progression
* No concurrent palliative radiotherapy
* See Disease Characteristics
* At least 4 weeks since prior major surgery
* No concurrent immunosuppressive drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2000-07; Primary Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Response rate using Response Evaluation Criteria in Solid Tumors (RECIST) | Up to 12 months
Toxicity assessed using Common Toxicity Criteria (CTC) version 2.0 | Up to 12 months

SECONDARY OUTCOMES:
Degree of NK cell expansion | Up to 12 months
Effectiveness of patients' PBMCs in a standard ADCC assay directed against HER2 target cells | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles Shapiro, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States